CLINICAL TRIAL: NCT00394017
Title: Implementation of an E-learning Program in Diagnostic Evaluation of Dementia by Reminders: A RCT Among General Practitioners in Copenhagen
Brief Title: The Use of Reminders in Implementing an E-learning Program in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Frans Boch Waldorff /MD PhD, Research Unit Of General Practice, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CPH-06-01-FEAP
Record Dates: First submitted 2006-10-26; First posted 2006-10-31 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Dementia
Keywords: Heading Health Plan Implementation; Computer-Assisted Instruction; General Practice; Dementia; education
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention group (Active Comparator): Reminder letters and usual implementations vs. usual implementation
  Interventions: Behavioral: Reminder letters
- Control group (No Intervention): usual implementations
  Interventions: Behavioral: Reminder letters

INTERVENTIONS:
Behavioral: Reminder letters — 3 mailed reminder letters

SUMMARY:
To evaluate General Practitioners use and reuptake of an e-learning programme in diagnostic evaluation of dementia after an intervention consisting of three mailed reminder letters.

There is no direct patient involvement in this study.

DETAILED DESCRIPTION:
The three mailed reminder letters will be mailed to the General Practitioners (GPs) in January 2007. The Periods where the e-learning programme will identify GPs using the programme are: Period before: November 1. and 6 weeks forward. Period after: Medio marts and 6 weeks forward.

All log files are kept anonymous for the principal study investigator by the Danish Medical Association.

ELIGIBILITY:
Inclusion Criteria:

* General Practitioners working in Copenhagen Municipality October 1st 2006

Exclusion Criteria:

* General Practitioners stopping to work in study period

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The proportion of General Practices using the e-learning programme at least once in periods monitored.

SECONDARY OUTCOMES:
The number of logins in the periods monitored.
The time og logins in the periods monitored.
The number of logins in working hours in the periods monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Frans B Waldorff, PhD, Principal Investigator — Research Unit of General Practice
Locations (1):
- Research Unit of General Practice, Copenhagen, Capital Province, Denmark